CLINICAL TRIAL: NCT07292363
Title: Evaluation of Inflammation-Related Endothelial Barrier Dysfunction in Patients With Chronic Apical Periodontitis Before and After Endodontic Treatment
Brief Title: Inflammation-Related Endothelial Barrier Dysfunction in Patients With Apical Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 0094485/II
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Apical Periodontitis; Healhty
Keywords: Endodontics; Apical Periodontitis; Inflammation; Endothelial barrier permeability
MeSH Terms: conditions — Periapical Periodontitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AP group: Healthy subjects with apical periodontitis between 25-55 years
  Interventions: Other: Apical lesions cure
- Control Group: Healthy subjects without apical periodontitis between 25-55 years

INTERVENTIONS:
Other: Apical lesions cure — Treatment of apical lesions
  Groups: AP group

SUMMARY:
Inflammation is a common factor in chronic periodontitis and systemic diseases. However, to date, there is no scientific evidence supporting a causal effect of inflammation caused by apical periodontitis on endothelial barrier dysfunction.

A case-control study was designed to evaluate serum levels of endothelial barrier dysfunction factors in a sample of healthy patients aged 25 to 55, with or without apical periodontitis, before endodontic treatment and 6 and 12 months after treatment.

The aim of this study is to investigate the potential relationship between the presence of chronic endodontic lesions and inflammation-related alterations of the endothelial barrier that may compromise its integrity, as well as to determine whether endodontic treatment can reduce these factors, thereby preventing changes in endothelial permeability.

DETAILED DESCRIPTION:
Systemically healthy, informed, and consenting patients of both sexes under 55 years of age with a diagnosis of apical periodontitis who undergo endodontic treatment will be enrolled as cases and monitored at 6 and 12 months after treatment. Systemically healthy, informed, and consenting patients of both sexes under 55 years of age without apical periodontitis will be enrolled as control subjects.

The study has been designed to assess serum levels of tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β), interleukin-6 (IL-6), and interleukin-8 (IL-8), as well as the endothelial junctional proteins zonula occludens-1 (ZO-1), claudin-5, and vascular endothelial cadherin (VE-cadherin), using enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* 25-55 years
* in general health
* with or without endodontic disease

Exclusion Criteria:

* under 25 years
* over 55 years
* subjects with systemic or oral diseases other than endodontic affections
* patients who underwent other dental treatments in the previous 6 months

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Dental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Quantification of serum inflammatory cytokines (TNF-α, IL-1β, IL-6 and IL-8) and endothelial integrity factors (ZO-1, Claudin-5 and VE-cadherin) by ELISA assays in healthy subjects and patients before endodontic treatment | Baseline serum levels dosage of evaluated factors in control group and AP group.
  Dosage of serum TNF-α, IL-1β, IL-6, IL-8 and ZO-1, Claudin-5 and VE-cadherin levels by ELISA assays measured as pg/ml of serum in healthy subjects and patients before endodontic treatment - baseline. Data relative to each evaluated serum protein will be aggregated as healthy (control group) versus pathological (AP group) individuals.
Quantification of serum inflammatory cytokines (TNF-α, IL-1β, IL-6 and IL-8) and endothelial integrity factors (ZO-1, Claudin-5 and VE-cadherin) by ELISA assays in healthy subjects and patients after 6 months of endodontic treatment | 6 months post-treatment serum levels dosage of evaluated factors in control group and AP group.
  Dosage of serum TNF-α, IL-1β, IL-6, IL-8 and ZO-1, Claudin-5 and VE-cadherin levels by ELISA assays measured as pg/ml of serum in healthy subjects and patients- 6 months post-treatment. Data relative to each evaluated serum protein will be aggregated as healthy (control group) versus pathological (AP group) individuals.
Quantification of serum inflammatory cytokines (TNF-α, IL-1β, IL-6 and IL-8) and endothelial integrity factors (ZO-1, Claudin-5 and VE-cadherin) by ELISA assays in healthy subjects and patients after 12 months of endodontic treatment | Time Frame: 12 months post-treatment serum levels dosage of evaluated factors in control group and AP group.
  Dosage of serum TNF-α, IL-1β, IL-6, IL-8 and ZO-1, Claudin-5 and VE-cadherin levels by ELISA assays measured as pg/ml of serum in healthy subjects and patients- 12 months post-treatment. Data relative to each evaluated serum protein will be aggregated as healthy (control group) versus pathological (AP group) individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Pasqualini, DDS Ass Prof, Principal Investigator — University of Turin, Department of Surgical Sciences - Dental School
Locations (2):
- Italy (2):
  - Department of Oncology - University of Turin, Turin, Italy
  - Endodontics, Department of Surgical Sciences - Univeristy of Turin, Turin, Italy